CLINICAL TRIAL: NCT03902093
Title: Longitudinal Study of External Auditory Canal Morphology With Regards to Extended-wear Hearing Instrument
Brief Title: Morphology Effects of Extended Wear Hearing Instrument
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is withdrawn due to no enrollment, due to COVID pandemic.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kristina Rousso, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-19-00205
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Hearing Loss
Keywords: hearing loss, hearing aid
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hearing Aid (Experimental): Actual Patients in the clinic will be evaluated by their Audiologist, if they are candidates to use the Lyric Hearing aid they will be asked if they want to participate in the study which will include imaging of the ear canal with a device similar to the regular ear device used in the clinic to check if there are any changes to the morphology of the ear canal.
  Interventions: Diagnostic Test: Morphology changes with extended wear hearing aid

INTERVENTIONS:
Diagnostic Test: Morphology changes with extended wear hearing aid — Possible changes in morphology due to wearing an extended wear hearing aid device will be assessed with imaging

SUMMARY:
The lyric hearing device is a commercially available device produced by Sonova, and designed to be used for extended periods of time. We further want to investigate the morphology of the tissue around the device at different periods of time after the device has been fitted and used for a while.

An initial imaging of the tissue will be taken for baseline measurements. Questionnaires will also be used to assess patients satisfaction with the device and cognitive abilities.

DETAILED DESCRIPTION:
If the person seems to be a good candidate for the study, the Audiologist could discuss with the patient the time involved in the study and arrange an appointment with the patient if interested.

A series of appointments are designed to follow up the patient's development with the device at determined times during the process. On the first appointment the patient will be consented prior to any tests or health services given.

The first and last appointments are the longest ones with a duration of about 1 and a half hours for questionnaires, medical history, and device fitting. Additionally, all appointments include measurement of ear canal relative humidity which should take a total of 30 minutes and imaging of the area to determine thickness and blood flow in the tissue surrounding the device. Follow-up appointments with the Audiologist will take 45 minutes for all basic procedures. The Lyric device is used commercially and Audiologist can provide it to patients already, but the purpose of this study is to use a pioneer technique with a device that looks inside the ear canal in the same way as a regular used speculum to look at details of the tissue around the device to see if any changes occur due to extended wear of the Lyric hearing aid device.

The complete study per person will be completed in about six months. An Audiologist will perform all the audiology testing plus the ear canal humidity measurements and his/her time will be covered by the sponsor (a total of 9 hours per patient). The Lyric devices will be provided on loan by the sponsor as well as the equipment and software needed to make the ear canal humidity measurements. The imaging measurements will be conducted by the Audiologist trained in using the handheld device.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in the USC Otolaryngology Clinic who are determined to be candidates for a Lyric extended wear hearing aid device by their treating Audiologist (in general people with mild to moderate hearing loss may be eligible).

Exclusion Criteria:

* Patients in the USC Clinic who are determined by the Audiologist not to be good candidates for the Hearing aid extended wear device (in general, people with severe hearing loss are not eligible).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Morphology imaging | Complete study will take about six months per person
  Imaging of the tissue at each appointment will be made

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Rousso, AuD, Principal Investigator — University of Southern California